CLINICAL TRIAL: NCT01974635
Title: Proprioception Testing in Persons With Sensorimotor Impairment
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device used for eye-blinks did not work as performed.
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Paul J. Cordo, Site Sub-Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 00009635
Record Dates: First submitted 2013-10-21; First posted 2013-11-01 (Estimated); Results first posted 2019-06-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Spinal Cord Injury; Stroke; Acquired Brain Injury
Keywords: Spinal Cord Injury; Robotic therapy; Rehabilitation; Sensation; Movement; Proprioception; Stroke; Acquired Brain Injury
MeSH Terms: conditions — Spinal Cord Injuries; Stroke; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AMES Therapy and Diagnostic (Experimental): During treatment, the AMES device rotates the hand, into flexion and extension, while the patient assists with this motion,and while the lengthening muscle(s) are vibrated mechanically. At the end of the treatment, several diagnostic tests are performed to measure the participant's level of proprioceptive perception. This study provides for 25 AMES treatments and diagnostic tests over 8-13 weeks, at a rate of 2-3 sessions per week.
  Interventions: Device: AMES Therapy

INTERVENTIONS:
Device: AMES Therapy — During the therapy session, the AMES device rotates the hand into flexion and extension, while the patient assists with this motion, as possible. At the same time, the AMES device provides sensory stimulation by vibrating the tendons of muscles stretched by the movement. The vibratory stimulus switches from one side of the limb to the other when the rotation reverses direction so that the sensory stimulation remains functionally related to the movement. The subject will receive visual bio-feedback of their contribution to the motor movement.

SUMMARY:
In this study, an FDA-cleared device and type of treatment called "AMES," which stands for Assisted Movement with Enhanced Sensation, will be used to determine whether sensation in the upper limb of individuals with incomplete spinal cord injuries, acquired brain injury, or stroke improves along with movement through treatment. We hypothesize that measureable improvement in the sensation of the upper limb will precede improvement in functional movement.

DETAILED DESCRIPTION:
The AMES device performs tests of sensorimotor impairment as well as delivering therapy. In this study, we are testing 2 additional diagnostic tests (i.e., Joint Position Test and "Frisbee" Test), both of proprioception, in order to determine which of the two is the best test of proprioception. Our hypotheses are: (1) both sensation and movement recover with AMES treatment, (2) sensory recovery precedes that of movement, (3) robotic delivery of the Joint Position Test produces more reliable test results than does manual delivery of this test, and (4) the Frisbee Test results will parallel those of the Joint Position Test.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic incomplete SCI, stroke or acquired brain injured ABI subjects.
* Able to tolerate sitting upright at for at least 1 hour.
* Significant, but not complete, motor deficit in the hand and wrist, as determined by the Study Physician performing the screening.
* Significant, but not complete somatosensory deficit in the hand and wrist as determined by the Study Physician performing the screening.
* Cognitively and behaviorally capable of complying with the regimen.

Exclusion Criteria:

* Fracture of the treated limb resulting in loss of range of motion.
* Progressive neurodegenerative disorder.
* DVT of the treated extremity.
* Uncontrolled seizure disorder.
* Uncontrolled high blood pressure/angina.
* Osteo- or rheumatoid arthritis limiting range of motion
* Contractures equal to or greater than 50% of the normal ROM.
* Chronic ITB therapy.
* Peripheral nerve injury of the treated extremity.
* Pain in affected limb or exercise intolerance.
* Participation in another therapy or activity-based program.
* Skin condition not tolerant of device.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Cordo, Ph.D, Study Director — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Cordo P, Lutsep H, Cordo L, Wright WG, Cacciatore T, Skoss R. Assisted movement with enhanced sensation (AMES): coupling motor and sensory to remediate motor deficits in chronic stroke patients. Neurorehabil Neural Repair. 2009 Jan;23(1):67-77. doi: 10.1177/1545968308317437. Epub 2008 Jul 21. PMID 18645190
- [Background] Backus D, Cordo P, Gillott A, Kandilakis C, Mori M, Raslan AM. Assisted movement with proprioceptive stimulation reduces impairment and restores function in incomplete spinal cord injury. Arch Phys Med Rehabil. 2014 Aug;95(8):1447-53. doi: 10.1016/j.apmr.2014.03.011. Epub 2014 Mar 28. PMID 24685386
- [Background] Cordo P, Wolf S, Lou JS, Bogey R, Stevenson M, Hayes J, Roth E. Treatment of severe hand impairment following stroke by combining assisted movement, muscle vibration, and biofeedback. J Neurol Phys Ther. 2013 Dec;37(4):194-203. doi: 10.1097/NPT.0000000000000023. PMID 24232364

RESULTS

PARTICIPANT FLOW:
Groups:
- AMES Therapy: The AMES device rotates the hand into flexion and extension, while the participant assists with this motion and receives visual feedback of the motion. At the same time, the AMES device vibrates the muscles stretched by the movement. The vibratory stimulus switches from one side of the limb to the other when the rotation reverses direction so. This study provides for 25 AMES training sessions over 8-13 weeks.
Period: Overall Study
Arm/Group | AMES Therapy
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- AMES Therapy: The AMES device rotates the hand into flexion and extension, while the participant assists with this motion and receives visual feedback of the motion. At the same time, the AMES device vibrates the muscles stretched by the movement. The vibratory stimulus switches from one side of the limb to the other when the rotation reverses direction so. This study provides for 25 AMES training sessions over 8-13 weeks. At the end of the intervention, the participant's proprioception (i.e., sense of joint position and movement) is tested by asking the participant, with eyes closed, to blink as the fingers and thumb or the wrist are rotated through a prescribed joint angle (i.e., target angle) by the AMES device.
Arm/Group | AMES Therapy
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Joint Position Test - AMES Device
Description: Testing proprioceptive sensation, the subject, with eyes closed, attempts to identify verbally the direction of motion (i.e., flexion or extension) as the AMES device randomly moves the subject's thumb and fingers, or the whole hand, into flexion and extension.
Time Frame: Immediately after each treatment on the AMES Device
Population: Device used for eye-blinks did not perform as expected. Study terminated prior to any further analyses.
Groups:
- AMES Therapy and Diagnostic: AMES therapy: During treatment, the AMES device rotates the hand, into flexion and extension, while the patient assists with this motion,and while the lengthening muscle(s) are vibrated mechanically. At the end of the treatment, several diagnostic tests are performed to measure the participant's level of proprioceptive perception. This study provides for 25 AMES treatments and diagnostic tests over 8-13 weeks, at a rate of 2-3 sessions per week.
  AMES Diagnostic: Immediately following the therapy session, the AMES device rotates the hand into flexion and extension, while the patient, with eyes closed, indicates verbally the perceived direction of motion.
Arm/Group | AMES Therapy and Diagnostic
Number analyzed (Participants) | 0

2. Secondary Outcome: Frisbee Test - Device
Description: Testing proprioceptive sensation, the AMES device moves the subject's wrist through a 30 degree range, at variable speeds, as the subject attempts to identify when their wrist reaches a particular target, either by opening contact between the thumb and index finger (if possible) or blinking the eyes. The subject receives feedback about the accuracy of the testing.
Time Frame: After each treatment on the AMES device.
Population: Eye-blink response device didn't perform as expected. Study terminated before any analysis performed.
Groups:
- AMES Therapy and Diagnostic: AMES therapy: During treatment, the AMES device rotates the hand, into flexion and extension, while the patient assists with this motion,and while the lengthening muscle(s) are vibrated mechanically. At the end of the treatment, several diagnostic tests are performed to measure the participant's level of proprioceptive perception. This study provides for 25 AMES treatments and diagnostic tests over 8-13 weeks, at a rate of 2-3 sessions per week.
  AMES Diagnostic: Immediately following the therapy session, the AMES device rotates the hand into flexion or extension, while the patient, with eyes closed, indicates the moment he/she perceives the hand passes through a prescribed joint angle.
Arm/Group | AMES Therapy and Diagnostic
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- AMES Therapy and Diagnostic: AMES therapy: During treatment, the AMES device rotates the hand, into flexion and extension, while the patient assists with this motion,and while the lengthening muscle(s) are vibrated mechanically. At the end of the treatment, several diagnostic tests are performed to measure the participant's level of proprioceptive perception. This study provides for 25 AMES treatments and diagnostic tests over 8-13 weeks, at a rate of 2-3 sessions per week.
  AMES Diagnostic: Either at baseline and 10-13 weeks later, or immediately following each therapy session, the participant performs a number of diagnostic tests to determine his/her level of proprioceptive perception.
Arm/Group | AMES Therapy and Diagnostic
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMES Therapy and Diagnostic (N=2)
Fall (Injury, poisoning and procedural complications) | 1 (1) — Participant fell at home. Not related to intervention or participation in study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes